CLINICAL TRIAL: NCT03312465
Title: Anatomical Shoulder™ Domelock System A Multicenter, Prospective and Retrospective, Non-Controlled Post-Market Clinical Follow-up Study
Brief Title: Anatomical Shoulder Domelock System Study
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2014-07E
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Avascular Necrosis; Revision Surgery; Conditions Consequent to Earlier Operations; Arthritis, Rheumatoid; Arthritis, Degenerative; Arthritis;Traumatic
Keywords: Total Shoulder Arthroplasty; Hemi Shoulder Arthroplasty
MeSH Terms: conditions — Osteonecrosis; Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AS Domelock System Subjects: Subjects that receive the Anatomical Shoulder Domelock System
  Interventions: Device: AS Domelock System

INTERVENTIONS:
Device: AS Domelock System — Hemi or Total Shoulder Arthroplasty

SUMMARY:
The objectives of this study are to confirm safety and performance of the Anatomical Shoulder Domelock System when used in hemi or total shoulder arthroplasty by analysis of standard scoring systems, radiographs and adverse event records.

DETAILED DESCRIPTION:
This study is a multicenter, prospective and retrospective, non-controlled PMCF study involving orthopaedic surgeons skilled in hemi and total shoulder arthroplasty procedures. A minimum of six study centers will be involved and a total number of 73 implants will be included into the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18-80 years of age, inclusive
* Patient is skeletally mature
* Patient is suffering from severe shoulder pain and disability requiring unilateral or bilateral HSA or TSA based on physical exam and medical history
* Patient has failed conservative treatment
* Patient meets at least one of the following indications:

  * Advanced wear and tear of the shoulder joint resulting from degenerative, posttraumatic or rheumatoid arthritis if bone stock is adequate.
  * Avascular necrosis
  * Conditions consequent to earlier operations
  * Optional use in revision: in some medical conditions (e.g., early revision when adequate bone stock exists), the surgeon may opt to use primary implants in a revision procedure.

Additional criteria for retrospective patients:

* patient has been implanted with the Domelock system before site initiation visit.
* information available must include at minimum demographic information, the operative report and details of the device implanted.

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program
* Patients who have any condition which would in the judgement of the Investigator place the patient at undue risk or interfere with the study. Any patient who is institutionalized, or is a known drug abuser, a known alcoholic or anyone who cannot understand what is required of them
* Patient is known to be pregnant or breastfeeding
* Patient meets at least one of the contraindications:

  * Patient's physical conditions that would impair adequate implant support and/or prevent the use of an appropriately sized implant, e.g., previous surgery, insufficient quality or quantity of bone, neuromuscular compromise or vascular deficiency in the affected limb in sufficient degree to endanger the success of the intervention e.g., absence of musculoligamentous supporting structures, joint neuropathy or other conditions that may lead to inadequate skeletal fixation
  * Signs of infection
  * Severe instability secondary to advanced loss of osteochondral structure
  * Charcot's shoulder (neuroarthropathy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from severe shoulder pain and disability indicated for implantation of the Anatomical Shoulder Domelock System in hemi or total shoulder arthroplasty and who meet all inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2032-12-09 (Estimated); Study Completion 2032-12-09 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship | 10 Years
  The primary endpoint of this study is defined by the survival of the implant at 10 years which is based on removal or intended removal of the prosthesis and will be determined using Kaplan Meier method.

SECONDARY OUTCOMES:
Clinical Performance | 5 Years
  The secondary endpoint is defined by the performance of the Anatomical Shoulder Domelock System at 5 years, which is assessed by the Constant and Murley score.
  The Constant and Murley score is a 100-point functional shoulder assessment tool in which higher scores reflect increased function. The subjective variables are pain (15 points) and function (activities of daily living - sleep, work, recreation/sport; 20 points), for a total of 35 points. The objective variables are active range of motion (clinician assessment; 40 points) and strength (25 points), for a total of 65 points.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet Clinical Operations
Locations (6):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Germany (2):
  - Krankenhaus Maria Hilf, Daun
  - HELIOS ENDO-Klinik Hamburg, Hamburg
- Switzerland (2):
  - Univeritätklinik Bagrist, Zurich, Canton of Zurich
  - Universitätsspital Basel, Basel
- Royal Derby Hospital, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No